CLINICAL TRIAL: NCT07126990
Title: Clinical Study of a Novel Oncolytic Virus Ad-TD-nsIL12 in the Treatment of Primary High-grade Glioma
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xiaorong Wu (Industry)
Collaborators: Beijing Bio-Targeting Therapeutics Technology Co., Ltd (Industry)
Responsible Party: Sponsor-Investigator, Xiaorong Wu, Sanbo Brain Hospital,Capital Medical University, Beijing Bio-Targeting Therapeutics Technology Co., Ltd
Organization: Beijing Bio-Targeting Therapeutics Technology Co., Ltd (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-01-107
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-08

CONDITIONS: Glioma
Keywords: To evaluate the effectiveness of new oncolytic adenovirus Ad-TD-nsIL12 in the treatment of patients with functional area and thalamic primary HGG
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment of patients with non-functional areas, functional areas and primary HGG of the thalamus (Experimental): Ommaya capsule was placed for intratumoral injection at a dose of 1x10^10vp
  Interventions: Biological: Novel oncolytic virus Ad-TD-nsIL12

INTERVENTIONS:
Biological: Novel oncolytic virus Ad-TD-nsIL12 — Ommaya capsule was placed for intratumoral injection at a dose of 1×10^10vp

SUMMARY:
Clinical study of a novel oncolytic virus Ad-TD-nsIL12 in the treatment of primary high-grade glioma

DETAILED DESCRIPTION:
This study will conduct two prospective, single-arm, single-center, exploratory clinical trials aimed at assessing the preliminary efficacy and safety of the novel oncolytic adenovirus Ad-TD-nsIL12 in treating primary HGG. Trial 1 will preliminarily evaluate the efficacy and safety of Ad-TD-nsIL12 as neoadjuvant treatment for patients with non-functional zone primary HGG; Trial 2 will preliminarily evaluate the efficacy and safety of Ad-TD-nsIL12 in treating patients with functional zone and thalamic primary HGG, as well as their quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years old (including cut-off value), both male and female;
2. Glioma that meets the 2021 edition of the World Health Organization (WHO) classification criteria for central nervous system tumors and has not undergone any anti-tumor treatment;
3. The lesion is located in the non-functional area (Experiment 1) / the lesion is located in the functional area and thalamus (Experiment 2);
4. Have an intracranial measurable target lesion (refer to the iRANO standard);
5. Karnofsky Performance Score (KPS) ≥ 60 points;
6. Expected survival ≥ 3 months;
7. Good organ function;
8. Subjects of childbearing potential and their partners who are sexually active must be willing to use a medically approved effective method of contraception, such as double-barrier contraception, during treatment and within 6 months after the last dose, and men agree not to donate sperm;
9. Women of childbearing potential, must have a negative blood pregnancy test result within 7 days before the first dose, and are willing to undergo additional pregnancy testing during the study. Females of childbearing potential who have not been surgically sterilized (i.e., bilateral tubal ligation, bilateral oophorectomy, or total hysterectomy) or who are not postmenopausal; Menopause is the cessation of menstruation for 12 months in women over 45 years of age ≥ and excludes other causes of amenorrhea. In addition, serum follicle-stimulating hormone (FSH) levels in women under 50 years of age must be in the postmenopausal range to confirm menopause.

Exclusion Criteria:

1. Received any anti-tumor therapy (referring to the tumor to be observed) in the past;
2. Underwent major organ surgery (excluding needle biopsy) or significant trauma within 4 weeks before the first dose, or required to undergo elective surgery during the study;
3. Known or suspected allergy to the active ingredients, excipients and contrast agents of the study drug;
4. Those with a history of organ transplantation or planned organ transplantation during the study;
5. Those with active infection or uncontrollable infection requiring intravenous systemic treatment, or unexplained fever >38.5°C during screening and before the first dose;
6. Severe coagulation disorders or other obvious evidence of bleeding risk; History of gastrointestinal bleeding; Any other ≥ CTCAE grade 2 bleeding event in the past 6 months;
7. Subjects who have received systemic steroid drugs (> 10 mg/day of prednisone or equivalent) or other immunosuppressive agents within 14 days before the first dose; The following are excluded: treatment with topical, ocular, intraarticular, intranasal, and inhaled corticosteroids; short-term use of corticosteroids for prophylactic treatment (e.g., to prevent contrast allergy);
8. Adverse reactions of previous anti-tumor therapy have not recovered to CTCAE 5.0 grade ≤ grade 1 (except for toxicities judged by the investigator to have no safety risk, such as alopecia, grade 2 peripheral neurotoxicity, etc.);
9. History of immunodeficiency, including positive HIV antibody test;
10. Active hepatitis B (HBsAg positive and HBV-DNA> 500 IU/ml or the lower limit of the test of the study center [only if the lower limit of detection of the study center is higher than 500 IU/ml]); Active hepatitis C (positive for HCV antibody and lower limit of HCV-RNA> detection by the study center), positive Treponema pallidum antibody;
11. Poorly controlled hypertension as judged by the investigator (arterial hypertension that is still uncontrolled under standard treatment: systolic blood pressure ≥160mmHg and/or diastolic blood pressure ≥100mmHg);
12. History of severe cardiovascular disease, such as: ventricular arrhythmia requiring clinical intervention; QTc interval> 480 ms; Acute coronary syndrome, congestive heart failure, stroke, or other grade III or above cardiovascular events within 6 months prior to the first dose; New York Heart Association (NYHA) cardiac function grade ≥ II or left ventricular ejection fraction (LVEF) < 50%;
13. Other uncured malignant tumors within or at the same time within the past 3 years, except for carcinoma in situ that is considered clinically curable, such as cervical cancer in situ and basal cell carcinoma of the skin;
14. Subjects with active or previously suffered autoimmune diseases that may recur (including but not limited to: systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc.), except for clinically stable autoimmune thyroiditis;
15. Those who have received live attenuated vaccines or recombinant vaccines within 4 weeks before the first dose, or inactivated vaccines within 2 weeks before the first dose;
16. Previous immunotherapy with irAE grade evaluation ≥3;
17. Those with two or more intracranial lesions, or extracranial metastasis;
18. Those with neoplastic lesions in the brainstem, cerebellum, posterior fossa or spinal cord, leptomeningeal disease;
19. Diffuse subependymal and subarachnoid disease;
20. Those with a history of encephalitis, multiple sclerosis, and other central nervous system infections;
21. Those with cerebral herniation syndrome;
22. Known alcohol or drug dependence;
23. Mental disorders or poor compliance;
24. Pregnant or lactating females;
25. The investigator believes that the subject has other serious systemic diseases or other reasons that are not suitable for participating in this clinical study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2028-08-30 (Estimated); Study Completion 2028-08-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effectiveness of new oncolytic adenovirus Ad-TD-nsIL12 in the treatment of patients with non-functional zones, functional zones and thalamic primary HGG | 12 months
  12-month survival rate (OS12): defined as the proportion of cases of subjects who are still alive from 12 months after receiving treatment with the virus to the total number of cases

CONTACTS AND LOCATIONS:
Locations (1):
- Sanbo Brain Hospital, Capital Medical University, Beijing, Haidian District, Beijing, Haidian District, China

IPD SHARING:
Plan to Share IPD: No